CLINICAL TRIAL: NCT05928156
Title: Blood Cancer Symptom Management App Randomized Controlled Trial
Brief Title: Multiple Myeloma/Chronic Lymphocytic Leukemia Coach RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00105025
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma; Chronic Lymphocytic Leukemia
Keywords: MM; CLL
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myeloma Coach or CLL Coach Mobile App (Experimental): Participants diagnosed with Multiple Myeloma will use the Myeloma Coach app and participants diagnosed with CLL (chronic lymphocytic leukemia) will use the the CLL Coach app. Pattern Health apps are built around "patterns" of scheduled activities. Users will encounter a list of activities to engage with for the day. There is also an option to complete activities in an ad hoc fashion.
  Interventions: Other: Myeloma Coach or CLL Coach Mobile App
- Springboard Beyond Cancer informational website (Placebo Comparator)
  Interventions: Other: Springboard Beyond Cancer informational website

INTERVENTIONS:
Other: Myeloma Coach or CLL Coach Mobile App — Symptom Tracking: Subjects will be asked to track their symptoms on a weekly basis, as well as given the opportunity to track these symptoms whenever they would like. Subjects will receive feedback tailored to their symptom severity with coaching on self management, including encouraging them to reach out to their health care team when symptoms are new, severe or increasing in severity. Subjects will also be able to look at graphs of symptom severity over time and share them with family and their health care team.
  Medication Adherence Reminders and Tracking, Activities - tools based on CBT (cognitive behavioral therapy) principles can be utilized at any time to manage emotional distress. Learn - information on cancer, its treatment, self managing physical and emotional symptoms, and supportive resources.
  Arms: Myeloma Coach or CLL Coach Mobile App
Other: Springboard Beyond Cancer informational website — Springboard Beyond Cancer (https://survivorship.cancer.gov) is designed to make it easy for those in treatment and post-treatment to access essential information to help them manage ongoing cancer-related symptoms, deal with stress, improve healthy behaviors, communicate better with healthcare teams, and seek support from friends and family.
  Arms: Springboard Beyond Cancer informational website

SUMMARY:
The purpose of this study is to test the effectiveness of evidence-informed mobile apps, Myeloma Coach and CLL Coach. These apps have been developed to help manage the physical and emotional symptoms experienced by multiple myeloma and chronic lymphocytic leukemia survivors. This study hopes to determine if a mobile app is a useful tool to help people manage commonly reported symptoms related to Multiple Myeloma (MM) and chronic lymphocytic leukemia (CLL).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Be a resident of the United States of America;
* Be able to read and write English
* Consistent access to the internet via a smartphone, tablet or computer
* Have a diagnosis of multiple myeloma or chronic lymphocytic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Change in Edmonton Symptom Assessment Scale (ESAS) | Baseline, 4 weeks, 8 weeks
  The ESAS is a validated 10 item survey index used to assessed symptoms. The total ranges from 0 to 60, with a higher score indicating higher physical symptom burden.
Change in NCCN Distress Thermometer | Baseline, 4 weeks, 8 weeks
  The NCCN Distress Thermometer (DT) is a one-item, 11-point Likert scale represented on a visual graphic of a thermometer that ranges from 0 (no distress) to 10 (extreme distress), with which patients indicate their level of distress over the course of the week prior to assessment.
Change in PROMIS (Patient-Reported Outcomes Measurement Information System) Short Form Global Health | Baseline, 4 weeks, 8 weeks
  This validated 10 item survey captures a person's self assessment of their global physical and global mental health. The possible score ranges from 0 to 20 points in each case. 0 points represent the patient's most severe physical and/or mental impairment, while 20 points represent the best possible state of health.
Change in severity of PTSD related symptoms as measured by PTSD Checklist (PCL5) | Baseline, 4 weeks, 8 weeks
  This validated 20 item measure has been used extensively in research. Scores consist of a total symptom severity score (from 0 to 80) from four subscales: Re-experiencing (items 1-5 - max score = 20), Avoidance (items 6-7 - max score = 8), Negative alterations in cognition and mood (items 8-14 - max score = 28), and Hyper-arousal (items 15-20 - max score = 24). Higher scores represent higher severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LeBlanc MR, LeBlanc TW, Yang Q, McLaughlin J, Irish K, Smith SK. A Mobile App to Support Self-Management in Patients with Multiple Myeloma or Chronic Lymphocytic Leukemia: Pilot Randomized Controlled Trial. JMIR Cancer. 2023 Jul 6;9:e44533. doi: 10.2196/44533. PMID 37410541